CLINICAL TRIAL: NCT00605358
Title: Increasing Use of Mental Health Services by Community Dwelling Adults With Depression
Brief Title: Increasing Use of Mental Health Services
Acronym: OpenDoor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Jo Anne Sirey, Associate Professor, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01MH079265-01A1 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Major Depression
Keywords: geriatric depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Door Intervention (Active Comparator): Subjects who receive the Open Door Intervention will work with the study counselor to identify barriers to participation in mental health treatment, set goals, and problem-solve, in addition to receiving a referral.
  Interventions: Behavioral: Open Door intervention
- Services Referral (No Intervention): Subjects who do not receive the Open Door intervention will receive:
  1. an evaluation
  2. referral to a local mental health provider
  3. booklet information on depression and mental health care, and will complete an application for HEAP, a Westchester County service that provides reduced rates from oil companies on heating to seniors.

INTERVENTIONS:
Behavioral: Open Door intervention — Open Door intervention subjects will:
  1. receive an evaluation
  2. receive a referral to a local mental health provider
  3. identify barriers, set goals and problem-solve to achieve a mental health evaluation using available resources.
  Other Names: West group
  Arms: Open Door Intervention

SUMMARY:
The purpose of this study is to test the effectiveness of Open Door (previously known as the Treatment Initiation Program [TIP]), a brief psychosocial intervention to address the psychological barriers to care and improve the use of mental health services by depressed community elderly. The intervention is designed to help the older adult identify the barriers, problem-solve to find solutions and mobilize the motivation to seek help. Open Door was developed to work collaboratively with an older adult who is depressed to improve access and adherence to mental health treatment.

DETAILED DESCRIPTION:
The primary aim of this research study did not change from the original application; it is to conduct a randomized controlled trial of the effectiveness of a brief, psychosocial intervention on engagement in mental health care among homebound depressed older adults. Engagement is defined as accepting a referral and attending a visit with a provider who could provide traditional mental health care (medication or psychotherapy). The intervention, now called Open Door, was developed to work collaboratively with an older adult who has depressive symptoms to address the barriers to care with the aim of helping them consider a referral and engage in mental health care. In prior research, this intervention has been found to improve treatment participation, reduce depressive symptoms and increase adherence to antidepressant therapy among depressed older adults in primary care and outpatient psychiatric settings. We propose that Open Door will improve the access to mental health care by reducing psychological barriers, providing education about care, and managing the resignation associated with the symptoms of depression among community dwelling depressed elders. Additionally, we believe that despite the heterogeneity of mental health care that may be received, Open Door will be associated with reduced depressive symptoms by empowering the older adult to initiate care for him/herself.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older
* Homebound
* Endorse depressive symptoms

Exclusion Criteria:

* Presence of significant alcohol or substance abuse or psychotic disorder
* High suicide risk, i.e. intent or plan to attempt suicide
* Cognitive impairment
* Inability to speak English
* Aphasia interfering with communication.
* Current use of antidepressants or psychotherapy

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2007-08; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Anne Sirey, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sirey JA, Bruce ML, Alexopoulos GS. The Treatment Initiation Program: an intervention to improve depression outcomes in older adults. Am J Psychiatry. 2005 Jan;162(1):184-6. doi: 10.1176/appi.ajp.162.1.184. PMID 15625220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older adults who were eligible for home-meals delivery were recruited into the study if they screened positive for depressive symptoms. Screens were completed by home meals staff, while all research interviews were completed by trained research assistants.
Pre-assignment Details: A number of participants were excluded from the trial after screening but prior to randomization, due to the following reasons:
  Non-English speaking, active suicidality, starting new antidepressant or therapy, cognitive impairment, substance abuse, psychosis.
Groups:
- Services Referral (Control): Subjects who do not receive the Open Door intervention will receive:
  1. an evaluation
  2. referral to a local mental health provider
  3. booklet information on depression and mental health care, and will complete an application for HEAP, a Westchester County service that provides reduced rates from oil companies on heating to seniors.
Period: Overall Study
Arm/Group | Open Door Intervention | Services Referral (Control)
Started | 81 | 80
Completed | 81 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Door Intervention | Services Referral (Control) | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 82.9 (9.0) | 81.0 (9.5) | 81.9 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 67 | 49 | 116
  Male | 14 | 31 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 75 | 73 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 17 | 25 | 42
  White | 64 | 53 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Engagement Defined as at Least One Visit With a Mental Health Provider Who Can Offer Treatment of Depression.
Description: Engagement was defined as at least one visit with a mental health provider, due to the fact that in some treatment settings, the initial evaluation and the onset of treatment both took place in the first visit.
  The primary outcome, engagement, was counted if the participant had engaged in mental health treatment by EITHER 12 weeks OR 24 weeks, based on research suggesting that older adults may take up to 6 months to follow through on a referral.
  Therefore, while there is only a single primary outcome (engaged or not), it could be fulfilled at either of the two follow-up time points, at 12 or 24 weeks.
Time Frame: 12 and 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Open Door Intervention | Services Referral (Control)
Number analyzed (Participants) | 81 | 80
percentage of participants | 74.1 | 56.3
Statistical Analysis 1: Comparison: Open Door Intervention vs Services Referral (Control); Participants in the Open Door Intervention and the Services Referral condition were compared on rates of engagement in mental health services over the study follow-up period; Test type: Superiority or Other; p = .018, Chi-squared; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.17 to 4.93]

ADVERSE EVENTS:
Time Frame: Adverse data were collected throughout the entire study period (three years).
Description: All participants were systematically asked if they had been hospitalized since the prior research visit. All participants were also assessed for depression and suicidality.
Arm/Group | Open Door Intervention | Services Referral (Control)
Serious Adverse Events (participants affected / at risk) | 14/81 | 17/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Open Door Intervention (N=81) | Services Referral (Control) (N=80)
Hospitalization (Injury, poisoning and procedural complications) | 9/20 (15) | 15/24 (16) — Hospitalizations occurred due to medical emergencies and falls
Active Suicidal Ideation (Psychiatric disorders) | 1 (1) | 2 (3)
Death (General disorders) | 4 (4) | 0 (0) — Death was either natural or expected, NOT related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No